CLINICAL TRIAL: NCT05984589
Title: A Prospective, Randomized, Controlled, Double-Arm Study of RISE (Re-Invent, Integrate, Strengthen, Expand) Personalized Self-Management Training (PSMT) Compared to Standardized Self-Management Training (SSMT) in Colorectal Cancer (CRC) Patients
Brief Title: Personalized Health Self-Management Training for Colorectal Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3C-24-9; 1K01HD110719 (NIH)
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Healthy Lifestyle; Behavior, Health; Health Behavior
Keywords: self-management training
MeSH Terms: conditions — Colorectal Neoplasms; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RISE-PSMT (Experimental): Personalized self-management training using RISE (Re-Invent, Integrate, Strengthen, Expand) program.
  Interventions: Behavioral: RISE Personalized Self-Management Training (PSMT)
- SSMT (Placebo Comparator): Standardized self-management training.
  Interventions: Behavioral: Standardized Self-Management Training (SSMT)

INTERVENTIONS:
Behavioral: RISE Personalized Self-Management Training (PSMT) — Along with patient education and internalization of self-determination, the RISE intervention focuses on replacing unhealthy habits with health-promoting habits. Ongoing practice and guidance in generating and enacting SMART (specific, measurable, achievable, realistic, and time-bound) health goals is the centerpiece of the RISE intervention. Working one-on-one with the PI, participants will set goals and develop practical strategies to establish sustainable healthy behavior (HB) change. Motivational interviewing, cognitive behavioral therapy, and patient education will accompany intensive collaborative problem-solving and creation of accountability structures to create lasting change. The 6-week intervention includes 2 in-person visits and 4 videoconference sessions.
  Arms: RISE-PSMT
Behavioral: Standardized Self-Management Training (SSMT) — Participants randomized to the control condition will receive 6 standardized sessions from one of the occupational therapy (OT) interveners, matched to the PSMT for setting. At these visits, participants will be presented with slides containing pre-specified, standardized didactic content about the World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) healthy behavior recommendations (HBRs). We hypothesize that these visits will control for the effect of research participation and increased knowledge about HBRs, and that simply providing standardized didactic content as an intervention modality without any personalization will have negligible effects on participants' healthy behaviors (HBs), self-efficacy, or quality of life. Content will follow the WCRF/AICR HBRs. Weeks 1-2 will focus on physical activity; weeks 3-4 will focus on diet and alcohol, and weeks 5-6 will focus on weight management and generalized strategies for HB change.
  Arms: SSMT

SUMMARY:
This is a Phase 2 prospective, randomized, controlled, double-arm study to assess personalized self-management training (PSMT) intervention efficacy and patient experiences compared to standardized self-management training (SSMT). A total of 120 colorectal cancer (CRC) patients will be enrolled and randomized 1:1 to complete a 6-week self-management training program (either PSMT or SSMT) to be carried out by licensed occupational therapists with doctoral training.

This study aims to examine whether PSMT is more effective in increasing adherence to healthy behavior recommendations compared to SSMT in CRC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of consent.
2. History of Stage I-IV colorectal cancer (CRC) within the past 5 years prior to enrollment.
3. Ability to speak, write, and read English sufficiently to allow for program participation.
4. Identified by self-report as having willingness and interest to work on at least one lifestyle-related risk factor. Lifestyle-related risk factors include diet, physical activity, body composition, alcohol use.
5. Scoring ≤3.5 on the World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) Health Behavior Adherence Scale or in the low-to-moderate range in any subcategory consistent with moderate to low adherence to healthy behavior recommendations (HBRs).
6. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Cognitive or mental impairments that in the opinion of the Principal Investigator or study physician would hinder the program participation.
2. Planning to have active anti-cancer treatment (including radiation, chemo, and/or major surgery) within 6 months after initial interventional or control session. Long-term hormonal/biologic therapy is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
To compare the difference in WCRF/AICR score between the intervention (RISE-PSMT) and control (SSMT) groups. | 12 weeks.
  Outcome measures contributing to each component of WCRF/AICR Healthy Behavior Adherence scale will be collected from baseline and end-of-study visits (Session 6 and Follow-up). The WCRF/AICR scale comprises of 7 categories with each category given a score for non-/low adherence, moderate/some adherence, or full adherence to each HBR. Total value ranges from 0 to 7 points, with a higher score indicating better adherence. HBR items include body composition, physical activity, diet, and alcohol use.

SECONDARY OUTCOMES:
The difference in general self-efficacy between the two groups after the 6-week self-management program will be measured by Patient-Reported Outcomes Measurement Systems (PROMIS) Item Bank v1.0 - General Self-Efficacy Short Form 4a. | 12 weeks.
  Responses to this questionnaire will be collected at Baseline (Session 1), End of Study Week 6 (Session 6), and Follow-up 6 Weeks Post-Session 6. The questionnaire asks the subject to rate their confidence levels in managing various situations, problems, and events. There are a total of 4 questions, and each question is answered on a scale of 1-4 where higher scores indicate the highest level of confidence. Total value ranges from 4 to 20, with a higher score indicating higher self-efficacy or highest level of confidence.
To evaluate the difference in health-related quality of life between the two groups after completion of the self-management program, we will use the PROMIS Scale v1.2 - Global Health questionnaire . | 12 weeks.
  Responses will be collected at Baseline (Session 1), End of Study Week 6 (Session 6), and Follow-up Visit (6 weeks post Session 6).The questionnaire includes the following components to assess subject's rating on their global physical and mental health: 6 questions are each answered on a scale of 1-5 where higher scores indicate excellent health, 1 question is answered on a scale of 1-5 where higher scores indicate being able to completely carry out everyday physical activities, and the last 3 questions are answered on a scale of 1-5 where higher scores indicate less frequency or no occurrences of fatigue, pain, or emotional problems.
To assess percent change across the various component scores on the WCRF/AICR (e.g. grams of fiber) to better understand what might be driving any changes in the overall WCRF/AICR composite score. | 12 weeks
  To assess percent change across the various component scores on the WCRF/AICR, the WCRF/AICR will be collected at Screening, Baseline (Session 1) unless screening visit was <30 days ago, End of Study Week 6 (Session 6), and Follow-up Visit (6 weeks Post Session 6).

CONTACTS AND LOCATIONS:
Overall Officials: Alix G Sleight, PhD, OTD, MPH, OTR/L, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Southern California, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No